CLINICAL TRIAL: NCT03543579
Title: An Observational Study of Cardiovascular Complications of Carfilzomib Treatment in Clinical Practice
Brief Title: Cardiovascular Complications of Carfilzomib Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Meletios A. Dimopoulos, Professor of Hematology, Department of Clinical Therapeutics National and Kapodistrian University of Athens, School of Medicine, Athens, Greece, University of Athens
Other Study IDs: 20168009
Record Dates: First submitted 2018-05-04; First posted 2018-06-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; Carfilzomib; Proteasome inhibition
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Peripheral blood mononuclear cells (PBMCs)
  * Red blood cells (RBCs)
  * Serum and plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multiple myeloma patients: Patients with multiple myeloma and an indication to receive carfilzomib

SUMMARY:
Accumulating evidence supports the hypothesis of a pathophysiological role of the Ubiquitin Proteasome System (UPS) in the process of atherosclerosis and vascular function. However the data are contradicting in respect to the direction of this association and therefore the net effect of UPS activity on the cardiovascular system is not known. Inhibitors of UPS are currently standard of care for patients with multiple myeloma (MM). Heart failure and hypertension have been reported in studies of carfilzomib, an irreversible 2nd generation proteasome inhibitor, both as a single agent and in combination with other drugs but their potential vascular toxicity is not adequately studied. Furthermore, as the role of the UPS has not been studied yet clinically but only in experimental and autopsy based studies, assessment of UPS inhibition in humans would facilitate understanding of the UPS-mediated pathophysiologic mechanisms in human atherosclerosis. Thus, this project may stimulate further research on the role of UPS in atherogenesis and potential new therapeutic approaches on vascular dysfunction may arise. We designed the following project in order to investigate the acute and chronic effect of Carfilzomib (CFZ) on cardiovascular function. Patients with an indication to receive CFZ will be recruited to be followed in the Clinical Therapeutics Department in pre-specified timepoints. Functional and structural measurements including markers of arterial stiffness and subclinical atherosclerosis will be performed using non-invasive well-validated techniques. Blood pressure will be also evaluated using 24h hour ambulatory monitoring. Evaluation of cardiac function will be performed at baseline and thereafter at 6 months or earlier if a suspicious event occurs necessitating evaluation of cardiac function. In parallel and at each time point, the activity of UPS and intracellular levels of ubiquitin conjugates will be measured in peripheral blood mononuclear cells (PBMCs) and red blood cells (RBCs) using enzymatic proteasome activity assays and western blot techniques, respectively.

DETAILED DESCRIPTION:
This is an observational, non interventional, prospective study. Patients with relapsed or refractory multiple myeloma who have received at least one prior line of therapy and who receive carfilzomib with dexamethasone according to the approved dose and schedule will be included in this observational study. No specific treatment intervention related to the study is going to be performed. No specific harms or benefits are expected due to study investigations.

Objectives and Purpose: The present study will assess patients with multiple myeloma receiving the proteasome inhibitor carfilzomib (CFZ), in order to investigate, in vivo, a wide spectrum of human atherosclerosis indices, from cardiovascular risk factors to subclinical atherosclerosis at multiple successive stages in a human model under conditions of global UPS inhibition, and correlate with cardiovascular complications associated with carfilzomib therapy, in patients receiving carfilzomib with dexamethasone.

Primary objective: To investigate cardiovascular complications and the role of the UPS inhibition on atheromatosis and vascular function and inflammation, in patients with relapsed or refractory myeloma who are receiving carfilzomib and dexamethasone.

Secondary objective(s): To outline the clinical significance of carfilzomib toxicity in hemodynamic parameters and vascular function and structure in humans

Duration of the study: Patients will receive therapy until disease progression or as per physician's decision regarding the patient's best interest and according to the approved indications. Study accrual and collection of data will be completed in two years. The study can be terminated for any reason and at any time by the Sponsor.

Population: The study will include patients with relapsed or refractory multiple myeloma who have received at least one prior line of therapy (2) and who according to physicians' decision are treated with carfilzomib dexamethasone in the approved indication, doses and schedule. Briefly, patients aged 18 years or older with relapsed or refractory multiple myeloma, Eastern Cooperative Oncology Group performance status of 0 to 2, at last one prior treatments, will be included.

Carfilzomib treatment: According to the approved indications patients will be given carfilzomib at a dose of 20 mg/m2 on days 1 and 2 of cycle 1; and thereafter at a dose of 56 mg/m2, in a 30 min intravenous infusion, on days 1,2,8,9,15 and 16. Dexamethasone (40mg IV) will be administered 24-48 hours before first CFZ infusion in order to assess the individual vascular effects of each drug separately; subsequently dexamethasone will be given IV at a dose of 20 mg on days 1,2,8,9,15 and 16, and orally on days 22 and 23 of a 28-day cycle. The rationale for using these doses is based on the results of the ENDEAVOR study and the approved indications and dosing of KYPROLIS. Intravenous hydration (250-500 mL before and after dose administration) is going to be given during cycle 1 and at the investigator's discretion thereafter.

Sample size: This is an observational study with non interventional design. Sample size calculation is made on the basis of previous data indicating that at least 2% absolute difference in Flow mediated dilatation (FMD) (corresponding to 20-30% relative difference) is considered significant and clinically relevant. With the null hypothesis being that CFZ/Dex therapy is associated with <10% relative difference in FMD and the alternative hypothesis being that a ≥30% difference is considered as significant, and with an a=0.05, a sample of 40 patients is required for 90% power of detecting these differences (all tests are 2-sided). A dropout rate of 15% is assumed. A total number of 46 patients is thus calculated to be enrolled.

Studied parameters History record: A detailed history will be obtained from every subject and all possible risk factors that could be associated with an increased risk of cardiac and vascular adverse events including thorough clinical examination along with ECG and cardiac echocardiography to ensure that every patient has an ejection fraction ≥40% thus being eligible for enrollment.

Assessment of arterial stiffness: Arterial stiffness in the aorta by measurement of pulse wave velocity (PWV).

Central blood pressures and reflected waves in the aorta: Non-invasive estimation of aortic pressure waveforms and reflected waves by pulse wave analysis (PWA) will be performed. The following indices are measured: a. augmentation index (AI, percentage) normalized for the heart rate of 75 bpm, expressed as a percentage of the aortic pulse pressure, b. central systolic and diastolic pressures (cBP), c. time to the beginning of the reflected wave (in milliseconds) and d. blood pressure amplification calculated as the ratio of peripheral pulse pressure: central pulse pressure.

Endothelial function by ultrasound measurement of endothelium-dependent flow-mediated dilatation (FMD): Endothelial function will be assessed by Flow Mediated Dilatation (FMD)

Carotid and Femoral Intima-Media Thickness (IMT): Carotid intima-media thickness (ccIMT) will be measured at the distal 1.0 cm of the common carotid proximal to the bifurcation. Femoral IMT (fIMT) will be measured on each side, scanning a 1cm-long arterial segment proximal to the femoral bifurcation, defined as the common femoral artery segment and the average value of IMT of the far wall will be estimated.

Ankle Brachial Index (ABI): The ABI is a simple, non-invasive diagnostic test for lower-extremity peripheral arterial disease (PAD) with high validity of the test for stenosis ≥50% in leg arteries (sensitivity ≈95% and specificity ≈100%).

All the above mentioned vascular measurements will be performed at each time point, that is on baseline and days 1,2,8,9,15 and 16 of cycle 1 and on days 1,2 of cycle 2 and 3 before and 2 hours after drug administration. The B-Mode ultrasound of the carotid and femoral arteries will only be performed at baseline. On cycle 6 all vascular measurements will be repeated to assess the chronic effect of proteasome inhibition on vascular function and atherosclerosis.

24-hour Ambulatory Blood Pressure Monitoring (ABPM): Patients will have their blood pressure monitored for 24 hours during the 1st day of cycles 1, 2, 3 and 6.

Cardiac Ultrasonography: Study participants will undergo a baseline echocardiographic examination before the initiation of the treatment.

Study of Proteasome activity: In order to examine the molecular and cellular effects of therapeutic inhibitors in blood cells of MM patients, we will proceed to isolation of Red Blood Cells (RBCs) and Peripheral Blood Mononuclear Cells (PBMCs). The blood samples which will be used in this research will be collected between specific time points of therapeutic proteasomal inhibitors administration. The first day of the treatment (no drug administration) will be used as a control time point.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age
* Voluntary written informed consent before performance of any study-related procedure
* Documented relapsed or refractory multiple myeloma in need of therapy, after at least one previous line of therapy for myeloma
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2
* Willingness and ability to participate in study procedures

Exclusion Criteria:

* Anti-myeloma treatment within 2 weeks prior to Cycle 1, Day 1
* Cumulative dose of corticosteroids greater than or equal to the equivalent of 140mg prednisone for ≥4 days or a dose of corticosteroids greater than or equal to the equivalent of 40 mg/day of dexamethasone for ≥4 days within the 2-week period prior to Cycle 1, Day 1
* Previous allogeneic stem cell transplant; or Autologous Stem Cell Transplantation (ASCT) within 12 weeks before Cycle 1, Day 1
* Clinical signs of meningeal involvement of multiple myeloma
* Clinically significant cardiac disease, including:

  1. Myocardial infarction within 6 months, or unstable or uncontrolled condition (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV)
  2. Cardiac arrhythmia (CTCAE Grade 2 or higher) or clinically significant ECG abnormalities
  3. ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec
* Known active hepatitis B, or C.
* Known HIV infection.
* Prior or concurrent malignancy, except for the following:

  1. Adequately treated basal cell or squamous cell skin cancer.
  2. Any cancer (other than in-situ) from which the subject has been disease-free for 3 years prior to study entry.
* Any of the following laboratory test results during Screening:

  1. Absolute neutrophil count ≤1.0 × 109/L;
  2. Hemoglobin level ≤7.5 g/dL (≤5 mmol/L);
  3. Platelet count <75 × 109/L in patients in whom <50% of bone marrow nucleated cells are plasma cells and <50x109/L in patients in whom more than 50% of bone marrow nucleated cells are plasma cells;
  4. Alanine aminotransferase level ≥2.5 times the upper limit of normal (ULN);
* Pregnant or nursing women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with relapsed or refractory multiple myeloma who have received at least one prior line of therapy and who according to physicians decision are treated with carfilzomib dexamethasone in the approved indication, doses and schedule. Briefly, patients aged 18 years or older with relapsed or refractory multiple myeloma, Eastern Cooperative Oncology Group performance status of 0 to 2, at last one prior treatments, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2017-03-23 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in endothelial function (Flow Mediated Dilatation in %) after drug administration | baseline and 24 hours
  FMD will be assessed with echo at specific timepoints and differences to baseline will be recorded

SECONDARY OUTCOMES:
Changes in carotid intima-media thickness (IMT) | baseline and 24 weeks
  Carotid IMT will be assessed at baseline and at the final time point.
Changes in LV Ejection fraction | baseline and 6 months
  Assessment of cardiac function with echo
  * low risk: baseline and 6 months
  * intermediate risk: baseline, 3 and 6 months
  * high risk: baseline, 1, 3 and months
Changes in systolic and diastolic strain and strain rate of LV | baseline and 6 months
  Assessment of cardiac function with echo

CONTACTS AND LOCATIONS:
Overall Officials: Efstathios Kastritis, Professor, Principal Investigator — Associate Professor of the Department of Clinical Therapeutics at the National and Kapodistrian University of Athens School of Medicine, Athens, Greece; Kimon Stamatelopoulos, Professor, Principal Investigator — Assistant Professor of the Department of Clinical Therapeutics at the National and Kapodistrian University of Athens School of Medicine, Athens, Greece
Locations (1):
- Department of Clinical Therapeutics, "Alexandra" General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li W, Garcia D, Cornell RF, Gailani D, Laubach J, Maglio ME, Richardson PG, Moslehi J. Cardiovascular and Thrombotic Complications of Novel Multiple Myeloma Therapies: A Review. JAMA Oncol. 2017 Jul 1;3(7):980-988. doi: 10.1001/jamaoncol.2016.3350. PMID 27632640
- [Background] Waxman AJ, Clasen S, Hwang WT, Garfall A, Vogl DT, Carver J, O'Quinn R, Cohen AD, Stadtmauer EA, Ky B, Weiss BM. Carfilzomib-Associated Cardiovascular Adverse Events: A Systematic Review and Meta-analysis. JAMA Oncol. 2018 Mar 8;4(3):e174519. doi: 10.1001/jamaoncol.2017.4519. Epub 2018 Mar 8. PMID 29285538
- [Background] Dimopoulos MA, Roussou M, Gavriatopoulou M, Psimenou E, Ziogas D, Eleutherakis-Papaiakovou E, Fotiou D, Migkou M, Kanellias N, Panagiotidis I, Ntalianis A, Papadopoulou E, Stamatelopoulos K, Manios E, Pamboukas C, Kontogiannis S, Terpos E, Kastritis E. Cardiac and renal complications of carfilzomib in patients with multiple myeloma. Blood Adv. 2017 Feb 27;1(7):449-454. doi: 10.1182/bloodadvances.2016003269. eCollection 2017 Feb 28. PMID 29296960
- [Background] Dimopoulos MA, Moreau P, Palumbo A, Joshua D, Pour L, Hajek R, Facon T, Ludwig H, Oriol A, Goldschmidt H, Rosinol L, Straub J, Suvorov A, Araujo C, Rimashevskaya E, Pika T, Gaidano G, Weisel K, Goranova-Marinova V, Schwarer A, Minuk L, Masszi T, Karamanesht I, Offidani M, Hungria V, Spencer A, Orlowski RZ, Gillenwater HH, Mohamed N, Feng S, Chng WJ; ENDEAVOR Investigators. Carfilzomib and dexamethasone versus bortezomib and dexamethasone for patients with relapsed or refractory multiple myeloma (ENDEAVOR): a randomised, phase 3, open-label, multicentre study. Lancet Oncol. 2016 Jan;17(1):27-38. doi: 10.1016/S1470-2045(15)00464-7. Epub 2015 Dec 5. PMID 26671818
- [Background] Morimoto RI, Cuervo AM. Proteostasis and the aging proteome in health and disease. J Gerontol A Biol Sci Med Sci. 2014 Jun;69 Suppl 1(Suppl 1):S33-8. doi: 10.1093/gerona/glu049. PMID 24833584
- [Background] Trougakos IP, Sesti F, Tsakiri E, Gorgoulis VG. Non-enzymatic post-translational protein modifications and proteostasis network deregulation in carcinogenesis. J Proteomics. 2013 Oct 30;92:274-98. doi: 10.1016/j.jprot.2013.02.024. Epub 2013 Mar 14. PMID 23500136
- [Background] Patterson C, Cyr D. Welcome to the machine: a cardiologist's introduction to protein folding and degradation. Circulation. 2002 Nov 19;106(21):2741-6. doi: 10.1161/01.cir.0000041145.30519.6b. No abstract available. PMID 12438302
- [Background] Palombella VJ, Rando OJ, Goldberg AL, Maniatis T. The ubiquitin-proteasome pathway is required for processing the NF-kappa B1 precursor protein and the activation of NF-kappa B. Cell. 1994 Sep 9;78(5):773-85. doi: 10.1016/s0092-8674(94)90482-0. PMID 8087845
- [Background] Herrmann J, Edwards WD, Holmes DR Jr, Shogren KL, Lerman LO, Ciechanover A, Lerman A. Increased ubiquitin immunoreactivity in unstable atherosclerotic plaques associated with acute coronary syndromes. J Am Coll Cardiol. 2002 Dec 4;40(11):1919-27. doi: 10.1016/s0735-1097(02)02564-0. PMID 12475450
- [Background] Versari D, Herrmann J, Gossl M, Mannheim D, Sattler K, Meyer FB, Lerman LO, Lerman A. Dysregulation of the ubiquitin-proteasome system in human carotid atherosclerosis. Arterioscler Thromb Vasc Biol. 2006 Sep;26(9):2132-9. doi: 10.1161/01.ATV.0000232501.08576.73. Epub 2006 Jun 15. PMID 16778122
- [Background] Herrmann J, Saguner AM, Versari D, Peterson TE, Chade A, Olson M, Lerman LO, Lerman A. Chronic proteasome inhibition contributes to coronary atherosclerosis. Circ Res. 2007 Oct 26;101(9):865-74. doi: 10.1161/CIRCRESAHA.107.152959. Epub 2007 Sep 6. PMID 17823377
- [Background] Stangl V, Lorenz M, Meiners S, Ludwig A, Bartsch C, Moobed M, Vietzke A, Kinkel HT, Baumann G, Stangl K. Long-term up-regulation of eNOS and improvement of endothelial function by inhibition of the ubiquitin-proteasome pathway. FASEB J. 2004 Feb;18(2):272-9. doi: 10.1096/fj.03-0054com. PMID 14769821
- [Background] Chade AR, Herrmann J, Zhu X, Krier JD, Lerman A, Lerman LO. Effects of proteasome inhibition on the kidney in experimental hypercholesterolemia. J Am Soc Nephrol. 2005 Apr;16(4):1005-12. doi: 10.1681/ASN.2004080674. Epub 2005 Feb 16. PMID 15716331
- [Background] Van Herck JL, De Meyer GR, Martinet W, Bult H, Vrints CJ, Herman AG. Proteasome inhibitor bortezomib promotes a rupture-prone plaque phenotype in ApoE-deficient mice. Basic Res Cardiol. 2010 Jan;105(1):39-50. doi: 10.1007/s00395-009-0054-y. Epub 2009 Aug 20. PMID 19693627
- [Background] Meiners S, Ludwig A, Lorenz M, Dreger H, Baumann G, Stangl V, Stangl K. Nontoxic proteasome inhibition activates a protective antioxidant defense response in endothelial cells. Free Radic Biol Med. 2006 Jun 15;40(12):2232-41. doi: 10.1016/j.freeradbiomed.2006.03.003. Epub 2006 Mar 31. PMID 16785037
- [Background] Ludwig A, Fechner M, Wilck N, Meiners S, Grimbo N, Baumann G, Stangl V, Stangl K. Potent anti-inflammatory effects of low-dose proteasome inhibition in the vascular system. J Mol Med (Berl). 2009 Aug;87(8):793-802. doi: 10.1007/s00109-009-0469-9. Epub 2009 Apr 28. PMID 19399470
- [Background] Meiners S, Ludwig A, Stangl V, Stangl K. Proteasome inhibitors: poisons and remedies. Med Res Rev. 2008 Mar;28(2):309-27. doi: 10.1002/med.20111. PMID 17880010
- [Background] Safar ME, Levy BI, Struijker-Boudier H. Current perspectives on arterial stiffness and pulse pressure in hypertension and cardiovascular diseases. Circulation. 2003 Jun 10;107(22):2864-9. doi: 10.1161/01.CIR.0000069826.36125.B4. No abstract available. PMID 12796414
- [Background] Mattace-Raso FU, van der Cammen TJ, Hofman A, van Popele NM, Bos ML, Schalekamp MA, Asmar R, Reneman RS, Hoeks AP, Breteler MM, Witteman JC. Arterial stiffness and risk of coronary heart disease and stroke: the Rotterdam Study. Circulation. 2006 Feb 7;113(5):657-63. doi: 10.1161/CIRCULATIONAHA.105.555235. PMID 16461838
- [Background] Van Bortel LM, Duprez D, Starmans-Kool MJ, Safar ME, Giannattasio C, Cockcroft J, Kaiser DR, Thuillez C. Clinical applications of arterial stiffness, Task Force III: recommendations for user procedures. Am J Hypertens. 2002 May;15(5):445-52. doi: 10.1016/s0895-7061(01)02326-3. PMID 12022247
- [Background] Papaioannou TG, Protogerou AD, Stamatelopoulos KS, Vavuranakis M, Stefanadis C. Non-invasive methods and techniques for central blood pressure estimation: procedures, validation, reproducibility and limitations. Curr Pharm Des. 2009;15(3):245-53. doi: 10.2174/138161209787354203. PMID 19149616
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Joannides R, Haefeli WE, Linder L, Richard V, Bakkali EH, Thuillez C, Luscher TF. Nitric oxide is responsible for flow-dependent dilatation of human peripheral conduit arteries in vivo. Circulation. 1995 Mar 1;91(5):1314-9. doi: 10.1161/01.cir.91.5.1314. PMID 7867167
- [Background] Chondrogianni N, Trougakos IP, Kletsas D, Chen QM, Gonos ES. Partial proteasome inhibition in human fibroblasts triggers accelerated M1 senescence or M2 crisis depending on p53 and Rb status. Aging Cell. 2008 Oct;7(5):717-32. doi: 10.1111/j.1474-9726.2008.00425.x. Epub 2008 Aug 1. PMID 18691182
- [Background] Tsakiri EN, Sykiotis GP, Papassideri IS, Gorgoulis VG, Bohmann D, Trougakos IP. Differential regulation of proteasome functionality in reproductive vs. somatic tissues of Drosophila during aging or oxidative stress. FASEB J. 2013 Jun;27(6):2407-20. doi: 10.1096/fj.12-221408. Epub 2013 Mar 1. PMID 23457214
- [Background] Tsakiri EN, Sykiotis GP, Papassideri IS, Terpos E, Dimopoulos MA, Gorgoulis VG, Bohmann D, Trougakos IP. Proteasome dysfunction in Drosophila signals to an Nrf2-dependent regulatory circuit aiming to restore proteostasis and prevent premature aging. Aging Cell. 2013 Oct;12(5):802-13. doi: 10.1111/acel.12111. Epub 2013 Jun 28. PMID 23738891